CLINICAL TRIAL: NCT06339437
Title: Enhanced Recovery After Surgery (ERAS) Protocol Does Early Implementation Improve The Outcome For Elective Laparoscopic Cholecystectomy Surgery
Brief Title: Enhanced Recovery After Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Ashiq, Principal Investigator, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Adeel3
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cholelithiases
Keywords: ERAS; GALL STONE DISEASE; LAPAROSCOPIC CHOLECYSTECTOMY
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Intervention Model Description: ERAS protocols applied
Who Masked: Outcomes Assessor
Masking Description: outcomeassessor was not told about group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): ERAS protocol applied in this group
  Interventions: Other: ERAS Protocol
- non ERAS group (No Intervention): conventional method of post op care was used

INTERVENTIONS:
Other: ERAS Protocol — Ehanced recovery after surgery protocols were applied
  Arms: ERAS group

SUMMARY:
this study will be conducted involving patients of all genders between the ages of 20 and 60 years who will undergo elective laparoscopic cholecystectomy for uncomplicated symptomatic gallstone disease. The study will be conducted in Department of West Surgical Ward, Mayo Hospital, Lahore, after receiving approval from the hospital's Ethical Committee. Patients having other co-morbid conditions, pregnant patients, and those undergoing laparoscopic cholecystectomy converted to open surgery will be excluded from the study. LFTs and other baseline investigations will be done routinely of every patient. Written informed consent will be obtained from all the patient. Patients will be divided into two groups with 30 patients in each group. Group A will consist of patient in whom ERAS protocol will be implemented and Group B in whom ERAS protocol will not be implemented.

DETAILED DESCRIPTION:
INTRODUCTION: Gallstone disease is most frequent gastrointestinal problems. Gallbladder stone formation can cause discomfort in the upper abdomen. The gallbladder is surgically removed by keyhole surgery, a process known as laparoscopic cholecystectomy, to address this problem. The enhanced recovery after surgery (ERAS) program applies evidence based perioperative interventions that, collectively, reduce morbidity and length of hospital stay METHODOLOGY: A study will be conducted involving patients of all genders between the ages of 20 and 60 years who will undergo elective laparoscopic cholecystectomy for uncomplicated symptomatic gallstone disease. The study will be conducted in Department of West Surgical Ward, Mayo Hospital, Lahore, after receiving approval from the hospital's Ethical Committee. Patients having other co-morbid conditions, pregnant patients, and those undergoing laparoscopic cholecystectomy converted to open surgery will be excluded from the study. LFTs and other baseline investigations will be done routinely of every patient. Written informed consent will be obtained from all the patient. Patients will be divided into two groups with 30 patients in each group. Group A will consist of patient in whom ERAS protocol will be implemented and Group B in whom ERAS protocol will not be implemented.

All patients were demonstrated about use of the VAS score. Duration of analgesia was recorded and additional requirement for analgesia was noted. Post-operative side effects i.e. nausea, vomiting, sedation and shivering were noted. Post-operative hospital stay was also noted. All data were noted and analyzed in to SPSS v25.0. Independent t-test was applied for the comparison of mean post-operative duration of analgesia and mean post-operative pain score between two groups taking p-value ≤0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

* • Ages between 20 to 60 years

  * All genders included
  * ASA class I and II
  * Undergoing elective laparoscopic cholecystectomy for uncomplicated symptomatic gallstone disease.

Exclusion Criteria:

* Patients having other co-morbid conditions like uncontrolled diabetes (BSR>300) and uncontrolled hypertension (Blood Pressure>180/110).
* Previous abdominal surgery documented previous medical records.
* Pregnant patients documented on history
* Those undergoing laparoscopic cholecystectomy converted to open surgery proved by per-operative findings
* Immunocompromised patients documented on previous medical records.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
PONV | 24 hours
  post op nausea and vomiting measured
Visual Analogue Scale score | 24 hours
  pain assessed by visual analogue scale and higher score means worse outcome and less score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Adeel A Gujjar, M.S, Principal Investigator — Consultant Surgeon
Locations (1):
- The Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
not sharing